CLINICAL TRIAL: NCT03892915
Title: Depression Care to Improve Adherence to Prevention of Mother-to-Child-Transmission (PMTCT) Care Continuum & Pregnancy Outcomes
Brief Title: Maternal Depression Treatment in HIV
Acronym: M-DEPTH
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: RAND (Other)
Collaborators: Makerere University (Other); Mildmay Uganda Limited (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-1041
Record Dates: First submitted 2019-03-21; First posted 2019-03-27 (Actual); Results first posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-09

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial with 4 sites randomly assigned to implement evidence-based depression care in addition to usual care and 4 sites randomly assigned to implement usual care only
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Depression Care (Experimental): Task-shifted depression care, consisting of (1) depression screening and psychoeducation, (2) depression diagnosis, and (3) evidence-based problem solving therapy (PST) or antidepressant therapy (ADT; for those with severe and refractory depression, or who decline PST), to be implemented by trained peer mothers and midwife nurses in addition to usual care.
  Interventions: Combination Product: evidence-based depression treatment
- Usual care (No Intervention): Usual care processes for treating depression consist of referrals to mental health specialists and access to the Family Support Group program (a nation wide Ministry of Health program for HIV+ women at public ANC clinics, consisting of monthly sessions designed to provide psychosocial support and education to promote pregnancy management and PMTCT adherence).

INTERVENTIONS:
Combination Product: evidence-based depression treatment — We will use a stepped care approach to depression treatment. Participants with clinical depression (defined as PHQ-9>9) will be offered either Problem Solving Therapy (PST) or Antidepressant Therapy (ADT), but those with moderate to moderately severe depression will be recommended PST, while those with severe depression will be recommended ADT. Participants with subthreshold depressive symptoms (PHQ-9: 5-9) will receive depression psychoeducation and continued depressive monitoring.
  Arms: Depression Care

SUMMARY:
Cluster randomized controlled trial to compare the effects of task-shifted, evidence-based depression care vs. usual care on adherence to each step of the prevention of mother-to-child-transmission (PMTCT) care cascade at 8 antenatal care (ANC) clinics in Uganda.

DETAILED DESCRIPTION:
This study is a cluster randomized controlled trial (RCT) to compare the effects of task-shifted, evidence-based depression care vs. usual care on adherence to each step of the PMTCT care cascade at 8 ANC clinics in Uganda. At 4 experimental sites, task-shifted, depression care will include (1) depression screening and psychoeducation, (2) depression diagnosis, and (3) provision of evidence-based problem solving therapy (PST), or antidepressant therapy (ADT) for those with severe and refractory depression (or who decline PST), to be implemented by trained peer mothers and midwife nurses, respectively. The 4 control sites will use usual care services for managing depression, which consist of referrals to a mental health specialist and access to the Family Support Group program (comprehensive, monthly multi-session psychosocial program to enhance pregnancy management and PMTCT adherence). At each site, 50 HIV-positive newly pregnant women (total n=400) who screen positive for potential depression will be enrolled and followed until 18-months post-delivery to assess how depression and depression alleviation relate to primary (adherence to each component of the PMTCT care continuum, maternal virologic suppression) and secondary (infant HIV status; post-natal maternal and child health outcomes) outcomes, as well as processes of depression care (treatment uptake and depression alleviation among clinically depressed patients). A cost-effectiveness analysis will be used to compare the two study arms.

ELIGIBILITY:
Inclusion Criteria:

* detection of pregnancy through 24 weeks gestation (to ensure at least 12 weeks remaining antenatal period for assessing adherence to all stages of PMTCT care cascade)
* HIV-positive
* positive screen for potential depression on 2-item Patient Health Questionnaire (PHQ-2>0)
* on ART for at least 4 weeks

Exclusion Criteria:

* unstable health (about to start ART or on ART < 4 weeks; active, untreated opportunistic infection)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 391 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2024-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Wagner, PhD, Principal Investigator — RAND
Locations (1):
- Makerere University, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
We will make the data publicly available in the form of an electronic database for researchers who successfully complete a registration process. Data will be de-identified. We will provide documentation in the form of a codebook in which each variable name and response options are defined. Users must agree to the conditions of use governing access to the public release data. Users must submit brief proposals regarding intended use of the data; the study team will determine the scientific soundness of the proposal, as well as whether adequate data protections in place, as part of the decision for the researcher to be able to access the public use dataset.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Following publication of the main paper(s) for this study and the grant end-date.
Access Criteria: Users must submit brief proposals regarding intended use of the data; the study team will determine the scientific soundness of the proposal, as well as whether adequate data protections in place, as part of the decision for the researcher to be able to access the public use dataset.

REFERENCES:
- [Derived] Wagner GJ, Ghosh-Dastidar B, Gwokyalya V, Faherty LJ, Beyeza-Kashesya J, Nakku J, Nabitaka LK, Akena D, Nakigudde J, Ngo V, McBain R, Lukwata H, Kyohangirwe L, Mukasa B, Wanyenze RK. Effects of M-DEPTH model of depression care on maternal depression, functioning, and HIV care adherence, and infant developmental over eighteen months post-partum: results from a cluster randomized controlled trial. BMC Pregnancy Childbirth. 2025 Apr 5;25(1):400. doi: 10.1186/s12884-025-07443-0. PMID 40188047
- [Derived] McBain R, Okunogbe A, Gwokyalya V, Wanyenze RK, Wagner G. Economic evaluation of Maternal Depression Treatment in HIV (M-DEPTH) for perinatal depression among women living with HIV in Uganda: a cost-effectiveness analysis. BMJ Public Health. 2024 Jul 16;2(1):e000754. doi: 10.1136/bmjph-2023-000754. eCollection 2024 Jun. PMID 40018208
- [Derived] McBain RK, Schuler MS, Rukundo T, Wanyenze RK, Wagner GJ. Trajectories of perinatal depression among women living with HIV in Uganda. J Glob Health. 2024 Sep 20;14:04147. doi: 10.7189/jogh.14.04147. PMID 39301593
- [Derived] Wagner GJ, Gwokyalya V, Faherty L, Akena D, Nakigudde J, Ngo V, McBain R, Ghosh-Dastidar B, Beyeza-Kashesya J, Nakku J, Kyohangirwe L, Nabitaka LK, Lukwata H, Mukasa B, Wanyenze RK. Effects of M-DEPTH Model of Depression Care on Maternal HIV Viral Suppression and Adherence to the PMTCT Care Continuum Among HIV-Infected Pregnant Women in Uganda: Results from a Cluster Randomized Controlled Trial at Pregnancy Completion. AIDS Behav. 2023 Sep;27(9):2902-2914. doi: 10.1007/s10461-023-04014-2. Epub 2023 Mar 13. PMID 36907945
- [Derived] Wagner GJ, Gwokyalya V, Akena D, Nakigudde J, McBain R, Faherty L, Ngo V, Nakku J, Kyohangirwe L, Banegura A, Beyeza-Kashesya J, Wanyenze RK. Stressors and Maladaptive Coping Mechanisms Associated with Elevated Perinatal Depressive Symptoms and Suicidality Among Women Living with HIV in Uganda. Int J Behav Med. 2023 Oct;30(5):743-752. doi: 10.1007/s12529-022-10124-3. Epub 2022 Sep 20. PMID 36127627
- [Derived] Wagner GJ, McBain RK, Akena D, Ngo V, Nakigudde J, Nakku J, Chemusto H, Beyeza-Kashesya J, Gwokyalya V, Faherty LJ, Kyohangirwe L, Nabitaka LK, Lukwata H, Linnemayr S, Ghosh-Dastidar B, Businge J, Mukasa B, Wanyenze RK. Maternal depression treatment in HIV (M-DEPTH): Study protocol for a cluster randomized controlled trial. Medicine (Baltimore). 2019 Jul;98(27):e16329. doi: 10.1097/MD.0000000000016329. PMID 31277180

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place between July 2019 and January 2021 at the antenatal clinic sites
Pre-assignment Details: Once enrolled, participants were automatically assigned to their group, given the cluster randomization (e.g., they received what their site was assigned to)
Units Other Than Participants: clinic site
Period: Overall Study
Arm/Group | Depression Care | Usual Care
Started | 191; 4 clinic site | 200; 4 clinic site
Completed | 171; 4 clinic site | 167; 4 clinic site
Not Completed | 20; 0 clinic site | 33; 0 clinic site
Not completed — Lost to Follow-up | 6 | 12
Not completed — Death | 0 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — unsuccessful delivery | 13 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Depression Care | Usual Care | Total
Number analyzed (Participants) | 191 | 200 | 391
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.3 (5.7) | 27.7 (6.2) | 27.5 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 191 | 200 | 391
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 191 | 200 | 391
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Uganda | 191 | 200 | 391
Any secondary education [Count of Participants; unit: Participants] | 79 | 61 | 140
In a committed relationship [Count of Participants; unit: Participants] | 154 | 168 | 322
Gestation week [Mean (Standard Deviation); unit: weeks] | 21.3 (6.4) | 21.4 (5.6) | 21.3 (6.0)
Newly diagnosed with HIV [Count of Participants; unit: Participants] | 41 | 40 | 81
undetectable HIV viral load [Count of Participants; unit: Participants] | 108 | 120 | 228
depressive symptoms [Mean (Standard Deviation); unit: units on a scale] — PHQ-9 (Patient Health Questionnaire, 9-item) total score (range is 0-27, with higher scores representing greater depression), measures depression
  units on a scale | 11.9 (4.5) | 13.6 (5.6) | 12.7 (5.2)

OUTCOME MEASURES:

1. Primary Outcome: Rate of Maternal HIV Viral Suppression
Description: Percentage of participants who achieve undetectable HIV viral load as measured by blood assay
Time Frame: Two months post pregnancy
Measure: Count of Participants; unit: Participants
Arm/Group | Depression Care | Usual Care
Number analyzed (Participants) | 191 | 200
Participants | 128 | 132
Statistical Analysis 1: Comparison: Depression Care vs Usual Care; Test type: Superiority; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.73 to 1.93]

2. Primary Outcome: Mean Maternal Antiretroviral (ART) Adherence
Description: Group mean percentage of prescribed ART doses taken as measured by pharmacy refill data
Time Frame: Past 6 months, assessed at 2 months after the completion of pregnancy
Measure: Mean (Standard Deviation); unit: percentage of prescribed doses taken
Arm/Group | Depression Care | Usual Care
Number analyzed (Participants) | 191 | 200
percentage of prescribed doses taken | 95.2 (15.4) | 90.8 (20.2)
Statistical Analysis 1: Comparison: Depression Care vs Usual Care; Test type: Superiority; beta coefficient = 5.33, Standard Error of Mean 5.39

3. Primary Outcome: Rate of Prevention of Mother-to-child-transmission (PMTCT) Care Retention
Description: Percentage of participants who continue to attend antenatal care (ANC) visits as measured by chart abstraction
Time Frame: through study completion, an average of 48 weeks
Population: Number of participants randomly assigned to this group
Measure: Count of Participants; unit: Participants
Arm/Group | Depression Care | Usual Care
Number analyzed (Participants) | 191 | 200
Participants | 184 | 185

4. Primary Outcome: Rate of Delivery in Health Facility
Description: Percentage of participants who delivery their baby of in a health facility as measured by chart abstraction
Time Frame: two months post pregnancy
Measure: Count of Participants; unit: Participants
Arm/Group | Depression Care | Usual Care
Number analyzed (Participants) | 191 | 200
Participants | 171 | 165
Statistical Analysis 1: Comparison: Depression Care vs Usual Care; Test type: Superiority; Odds Ratio (OR) = 1.85, 95% CI 2-sided [0.53 to 6.50]

5. Primary Outcome: Rate of Infant Use of ART
Description: Percentage of delivered infants who receive ART as measured by chart abstraction
Time Frame: First 6 weeks of life
Measure: Count of Participants; unit: Participants
Arm/Group | Depression Care | Usual Care
Number analyzed (Participants) | 191 | 200
Participants | 174 | 164
Statistical Analysis 1: Comparison: Depression Care vs Usual Care; Test type: Superiority; Odds Ratio (OR) = 2.73, 95% CI 2-sided [0.45 to 16.64]

6. Secondary Outcome: Depression Status
Description: Depression was assessed with the 9-item Patient Health Questionnaire (PHQ-9); total score range is 0-27, with higher scores representing greater depression. total score > 9 represents clinical depression and the binary depression status variable = yes (depressed).
Time Frame: 2 months postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Depression Care | Usual Care
Number analyzed (Participants) | 191 | 200
Participants | 37 | 102
Statistical Analysis 1: Comparison: Depression Care vs Usual Care; Test type: Superiority; Odds Ratio (OR) = 0.20, 95% CI 2-sided [0.05 to 0.83]

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Depression Care | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/191 | 2/200
Serious Adverse Events (participants affected / at risk) | 13/191 | 18/200
Other Adverse Events (participants affected / at risk) | 0/191 | 0/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Depression Care (N=191) | Usual Care (N=200)
death to fetus/newborn (Pregnancy, puerperium and perinatal conditions) | 13 | 18 — miscarriage, abortion, stillbirth, neonatal death

LIMITATIONS AND CAVEATS:
With all participants being stable on ART and exhibiting a consistent HIV/ANC care retention throughout the study, as well as most having an undetectable HIV viral load at baseline, this may have contributed to a ceiling effect and limited the generalizability of our findings. The benefits of depression care may be more evident among women with a greater range of engagement in care, which in turn may be related to increased vulnerability to post-partum depression.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-16): https://cdn.clinicaltrials.gov/large-docs/15/NCT03892915/Prot_SAP_000.pdf